CLINICAL TRIAL: NCT03507036
Title: Pilot Study: Clinical Assessment of Bipolar Radiofrequency Microneedling for Improved Laxity and Wrinkles of the Suprapatellar Skin
Brief Title: Radio Frequency Microneedling for Suprapatellar Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey M. Kenkel, Betty and Warren Woodward Chair in Plastic and Reconstructive Surgery, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 082017-079
Record Dates: First submitted 2017-10-26; First posted 2018-04-24 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Skin Laxity
Keywords: knee area; suprapatellar skin; aging; laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): All patients will undergo treatment with Profound system device. Using the radiofrequency and temperature setting within the FDA approved limits (460 +/- 5kHz and 65-75°C +/- 1°C), patients will be treated one time over the entire suprapatellar region bilaterally and followed for a 6 month period. The acute effect of the radiofrequency application will be determined by subjective and objective analysis using standard, close-up, 3D, cross-polarized, high resolution ultrasound, optical coherence tomography, transepidermal water loss measurements, and/or BTC 2000 measurements.
  Biopsies will be taken using 0.33mm WellTech Rapid Core 0.33mm Biopsy Punch. Biopsies will allow investigators to correlate changes seen in skin measurements with histology and gene expression.
  Interventions: Device: Profound system

INTERVENTIONS:
Device: Profound system — Profound system is a bipolar fractional radiofrequency device which uses microneedles and thermal heat to stimulate neocollagenesis. Based on the its effect on facial skin, it can be hypothesized that bipolar fractional radiofrequency will stimulate similar effect on suprapatellar skin, lifting and reducing laxity of the skin in that region. Bilateral suprapatellar regions will be identified and marked for treatment.

SUMMARY:
The human skin aging process is characterized by thinning dermis, atrophy of the extracellular matrix, and reduced collagen synthesis. Loss of collagen in the dermis is of aesthetic concern, as it is the main structural support in the dermis and its loss results in skin laxity. Photo-damaged skin, mostly due to UVR, causes degradation of elastic fibers. This is histologically seen as disorganized tangles of elastin. Additionally, as humans age, skin tends to appear more dry due to its poor hydration and turgor capacity. The use of minimally invasive aesthetic treatments in reducing signs of aging has been gaining in popularity over surgical treatments in recent years. Several energy types including, laser, radiofrequency, infrared, and ultrasound, have been developed for facial rejuvenation. These treatments induce controlled thermal damage into the dermis and cause collagen contraction and neocollagenesis resulting in skin tightening over several months. For improving appearance of other anatomical areas, micro-focused ultrasound has been the preferred method, but has shown limited success in tightening the suprapatellar skin.

As with facial skin aging, the suprapatellar skin loses elasticity with age and begins to sag. Noninvasive treatments used for the face may also be used in other anatomical areas to produce the same effects of tightening. Minimally invasive bipolar radiofrequency produces a controlled thermal injury in a fractional manner without damaging the dermal-epidermal junction, epidermis or subcutis. Radiofrequency, unlike lasers, are chromophore-independent providing better penetration than lasers, and spare sweat glands, sebaceous glands, and hair follicles.

DETAILED DESCRIPTION:
The Profound System is a bipolar fractional radiofrequency device which uses microneedles and thermal heat to stimulate neocollagenesis. Based on the its effect on facial skin, it can be hypothesized that bipolar fractional radiofrequency will stimulate similar effect on suprapatellar skin, lifting and reducing laxity of the skin in that region.

This study intends to evaluate the effectiveness of the Profound System on suprapatellar skin, which has been FDA approved for treatment of facial wrinkles and improvement in the appearance of cellulite. This device is a well studied and frequently used on facial skin, however, there are no studies showing its effectiveness elsewhere on the body.

There are alternative treatments that have been shown to decrease laxity of the suprapatellar skin, however, the studies include a small and limited population, and have not produced the desired effects in practice. The Profound device may be able to produce clinically significant improvement in laxity of the suprapatellar skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults between ages 18-75 years of age.
* Subjects who can read, understand, and sign the Informed Consent Form.
* Subjects willing and able to comply with all study requirements
* Fitzpatrick skin type I-III

Exclusion Criteria:

* Subjects with active localized or systemic infections.
* Immunocompromised subjects.
* Subjects with coagulation disorder.
* History of skin photosensitivity disorders, or use of photosensitizing drugs (e.g., tetracycline or sulfa drugs).
* Pregnant and/or lactating (All female volunteers will be advised about using birth control during the period of study).
* In the opinion of the trained clinician, subject is unwilling or unable to adhere to all study requirements, including application and follow-up visits.
* Subjects with a history of radiation therapy to the treatment area.
* Subject has a history of allergy to lidocaine or ester-based local anesthetics.
* Subjects with any skin pathology or condition that could interfere with evaluation or with the use of typical ancillary medical treatments or care used before, during or after treatments.
* Subjects have undergone dermatological procedures (e.g., laser or light treatments) for the treatment of wrinkles, skin resurfacing, or skin rejuvenation in the treatment area within 1 year of study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, MD, Principal Investigator — Chair & Professor
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tobin DJ. Introduction to skin aging. J Tissue Viability. 2017 Feb;26(1):37-46. doi: 10.1016/j.jtv.2016.03.002. Epub 2016 Mar 14. PMID 27020864
- [Background] Hantash BM, Ubeid AA, Chang H, Kafi R, Renton B. Bipolar fractional radiofrequency treatment induces neoelastogenesis and neocollagenesis. Lasers Surg Med. 2009 Jan;41(1):1-9. doi: 10.1002/lsm.20731. PMID 19143021
- [Background] Alster TS, Tanzi EL. Noninvasive lifting of arm, thigh, and knee skin with transcutaneous intense focused ultrasound. Dermatol Surg. 2012 May;38(5):754-9. doi: 10.1111/j.1524-4725.2012.02338.x. Epub 2012 Jan 23. PMID 22268509
- [Background] Alexiades-Armenakas M, Newman J, Willey A, Kilmer S, Goldberg D, Garden J, Berman D, Stridde B, Renton B, Berube D, Hantash BM. Prospective multicenter clinical trial of a minimally invasive temperature-controlled bipolar fractional radiofrequency system for rhytid and laxity treatment. Dermatol Surg. 2013 Feb;39(2):263-73. doi: 10.1111/dsu.12065. Epub 2012 Dec 28. PMID 23278964
- [Background] Gold M, Taylor M, Rothaus K, Tanaka Y. Non-insulated smooth motion, micro-needles RF fractional treatment for wrinkle reduction and lifting of the lower face: International study. Lasers Surg Med. 2016 Oct;48(8):727-733. doi: 10.1002/lsm.22546. Epub 2016 Aug 4. PMID 27490716

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: All patients will undergo treatment with Profound system device (bipolar fractional radiofrequency device which uses microneedles and thermal heat to stimulate neocollagenesis). Using the radiofrequency and temperature setting within the FDA approved limits (460 +/- 5kHz and 65-75°C +/- 1°C), patients will be treated one time over the entire suprapatellar region bilaterally and followed for a 6 month period. The acute effect of the radiofrequency application will be determined by subjective and objective analysis using standard, close-up, 3D, cross-polarized, high resolution ultrasound, optical coherence tomography, transepidermal water loss measurements, and/or BTC 2000 measurements.
  Biopsies will be taken using 0.33mm WellTech Rapid Core 0.33mm Biopsy Punch. Biopsies will allow investigators to correlate changes seen in skin measurements with histology and gene expression.
Period: Overall Study
Arm/Group | Treatment
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Photographic Knee Laxity and Texture Evaluation
Description: Photographs will be used to evaluate efficacy of treatment. The photographs from final visit will be compared to their baseline photographs and visually evaluated by the study team. The study team will assess the laxity from baseline to 6 months.
Time Frame: baseline and 6 months
Population: Reviewers were asked to evaluate the visible change in texture and laxity on a scale of 1-3. Worsened (1), No Change (2) and Improved (3).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 15
score on a scale
  Texture | 1.87 (0.52)
  Laxity | 2.02 (0.52)

2. Primary Outcome: Epidermal Thickness
Description: Skin Elasticity will be measured via BTC2000 prior to treatment (baseline), 7 days, 3 weeks, 3 months and 6 months post treatment. The change from baseline was calculated at each time frame.
Time Frame: baseline, 7 Days, 3 Weeks, 3 Months and 6 Months
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Treatment: All patients will undergo treatment with Profound system device on both knees using the radiofrequency and temperature setting within the FDA approved limits (460 +/- 5kHz and 65-75°C +/- 1°C). All subjects will be treated one time over the entire suprapatellar region bilaterally and followed for a 6 month period.
Arm/Group | Treatment
Number analyzed (Participants) | 15
mm
  Baseline | 96.53333 (10.2578)
  7 Days | 106.9 (24.0632)
  3 Weeks | 98.33333 (16.3524)
  3 Months | 92.36667 (9.55739)
  6 Months | 91.36667 (12.1414)

3. Primary Outcome: Dermal Thickness
Description: Dermal thickness will be masured via high resolution ultrasound prior to treatment (baseline), 7 days, 3 weeks, 3 months and 6 months post treatment. The change from baseline was calculated at each time frame.
Time Frame: Baseline, 7 Days, 3 Weeks, 3 Months and 6 Months
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Treatment: All patients will undergo treatment with Profound system device n both knees. Using the radiofrequency and temperature setting within the FDA approved limits (460 +/- 5kHz and 65-75°C +/- 1°C), patients will be treated one time over the entire suprapatellar region bilaterally and followed for a 6 month period.
Arm/Group | Treatment
Number analyzed (Participants) | 15
mm
  Baseline | 1104.7 (192.626)
  Day 7 | 1179.2 (177.83)
  Week 3 | 1241.367 (191.049)
  Month 3 | 1167.933 (150.659)
  Month 6 | 1122.233 (200.07)

4. Primary Outcome: Change in Blood Flow at 0.25mm
Description: Blood Flow will be measured via optical coherence tomography prior to treatment (baseline), 7 days, 3 weeks, 3 months and 6 months post treatment.
Time Frame: Baseline, Day 7, Week 3 Month 3 and Month 6
Population: Results at each visit show the change from baseline values.
Measure: Mean (Standard Deviation); unit: mm/s
Arm/Group | Treatment
Number analyzed (Participants) | 15
mm/s
  Baseline | 0.3294 (0.009815)
  Day 7 | 0.23 (0.41)
  Week 3 | -0.02 (0.37)
  Month 3 | 0.080534 (0.33661)
  Month 6 | 0.1045 (0.3411)

5. Primary Outcome: Transepidermal Water Loss
Description: Transepidermal Water Loss will be masured via Aquaflux prior to treatment (baseline), 7 days, 3 weeks, 3 months and 6 months post treatment. The change from baseline was calculated at each time frame.
Time Frame: Baseline, Day 7, Week 3, Month 3 and Month 6
Measure: Mean (Standard Deviation); unit: g/(m2h)
Arm/Group | Treatment
Number analyzed (Participants) | 15
g/(m2h)
  Baseline | 9.379 (2.05288)
  Day 7 | 9.6007 (2.1681)
  Week 3 | 10.9986 (3.9201)
  Month 3 | 11.744 (8.7825)
  Month 6 | 8.772 (1.966)

6. Primary Outcome: Skin Elasticity
Description: as for outcome 2
Time Frame: Baseline, Day 7, Week 3, Months 3 and Months 6
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Treatment: All patients will undergo treatment with Profound system device. Using the radiofrequency and temperature setting within the FDA approved limits (460 +/- 5kHz and 65-75°C +/- 1°C), patients will be treated one time over the entire suprapatellar region bilaterally and followed for a 6 month period. The acute effect of the radiofrequency application will be determined by subjective and objective analysis using standard, close-up, 3D, cross-polarized, high resolution ultrasound, optical coherence tomography, transepidermal water loss measurements, and/or BTC 2000 measurements.
  Biopsies will be taken using 0.33mm WellTech Rapid Core 0.33mm Biopsy Punch. Biopsies will allow investigators to correlate changes seen in skin measurements with histology and gene expression. that b
Arm/Group | Treatment
Number analyzed (Participants) | 15
mm
  Baseline | 0.80199 (0.1263)
  Day 7 | 0.811731094 (0.256170747)
  Week 3 | 0.82434 (0.1549)
  Month 3 | 0.77234 (0.11494)
  Month 6 | 0.74615 (0.11275)

7. Primary Outcome: Change in Skin Laxity
Description: BTC2000 will be used to measure skin laxity prior to treatment and post treatment. The BTC2000 is a non-invasive device that measures skin laxity by creating a negative pressure against the skin and calculates laxity when the pressure is released.
Time Frame: baseline, 7 days, 3 weeks, 3 months and 6 months
Population: Results at each visit show the change from baseline values.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment
Number analyzed (Participants) | 15
mm
  Baseline | 0.7408 (0.1200845)
  Day 7 | 12.5364 (27.762)
  Week 3 | 3.75791 (21.921)
  Month 3 | 0.85623 (21.253)
  Month 6 | -5.54778 (16.383)

8. Primary Outcome: Histological Analysis- Collagen 1
Description: Relative changes in protein abundance in biopsies taken at post treatment compare to control or entreated group will be quantified using an image processing software based on fluorescence signal intensity. The change from baseline was calculated at each time frame.
Time Frame: Baseline. Day 7 and 3 Months
Measure: Mean (Standard Deviation); unit: fluorescence intensity
Arm/Group | Treatment
Number analyzed (Participants) | 15
fluorescence intensity
  Baseline | 1.38 (0.51)
  Day 7 | 1.00 (0.23)
  Month 3 | 1.04 (0.23)

9. Primary Outcome: Gene Expression- Collagen 1
Description: Biopsies of the treated are will be taken prior to treatment and post treatment for gene expression analysis. This analysis will identify gene expression related to collagen formation and increased cell turnover. Fold change was calculated at each time point past baseline.
  Fold change = sample/average of the baseline.
Time Frame: Day 7, Month 3
Population: Results at each visit show the change from baseline values.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Treatment
Number analyzed (Participants) | 15
fold change
  Day 7 | 1.91 (1.68)
  Month 3 | 1.38 (0.57)

10. Primary Outcome: Epidermal Density
Description: Epidermal thickness will be masured via high resolution ultrasound prior to treatment (baseline), 7 days, 3 weeks, 3 months and 6 months post treatment. The change from baseline was calculated at each time frame.
Time Frame: Baseline, Day 7, Week 3, Month 3 and Month 6
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Treatment
Number analyzed (Participants) | 15
um
  Baseline | 0.00380558 (0.000635)
  Day 7 | 0.028518 (0.09374)
  Week 3 | 0.004336 (0.00232)
  Month 3 | 0.020107 (0.08714)
  Month 6 | 0.00392152 (2.783)

11. Primary Outcome: Histological Analysis- Collagen 3
Description: Relative changes in protein abundance in biopsies taken at post treatment compare to control or entreated group will be quantified using an image processing software based on fluorescence signal intensity. The change from baseline was calculated at each time frame. Sample/Average of the baseline.
Time Frame: Baseline, Day 7, Month 3
Population: Results at each visit show the change from baseline values.
Measure: Mean (Standard Deviation); unit: fluorescence intensity
Arm/Group | Treatment
Number analyzed (Participants) | 15
fluorescence intensity
  Baseline | 0.63 (0.17)
  Day 7 | 0.72 (0.18)
  Month 3 | 0.71 (0.28)

12. Primary Outcome: Histological Analysis- Elastin
Description: Relative changes in protein abundance in biopsies taken at post treatment compare to control or entreated group will be quantified using an image processing software based on fluorescence signal intensity. The change from baseline was calculated at each time frame. Samples/Average of the baseline
Time Frame: Baseline, Day 7, Month 3
Population: Results at each visit show the change from baseline values.
Measure: Mean (Standard Deviation); unit: fluorescence intensity
Arm/Group | Treatment
Number analyzed (Participants) | 15
fluorescence intensity
  Baseline | 1.29 (0.24)
  Day 7 | 0.90 (0.50)
  Month 3 | 0.58 (0.17)

13. Primary Outcome: Gene Expression- Collagen 3
Description: Biopsies of the treated are will be taken prior to treatment and post treatment for gene expression analysis. This analysis will identify gene expression related to collagen formation and increased cell turnover.
  Fold change = sample/average of the baseline.
Time Frame: Day 7, Month 3
Population: Results at each visit show the change from baseline values.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Treatment
Number analyzed (Participants) | 15
fold change
  Day 7 | 2.07 (1.68)
  Month 3 | 1.36 (0.96)

14. Primary Outcome: Gene Expression- Elastin
Description: as for outcome 13
Time Frame: Day 7, Month 3
Population: Results at each visit show the change from baseline values.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Treatment
Number analyzed (Participants) | 15
fold change
  Day 7 | 0.89 (0.41)
  Month 3 | 1.74 (1.37)

15. Primary Outcome: Gene Expression- Interluekin 6
Description: as for outcome 13
Time Frame: Day 7, Month 3
Population: Results at each visit show the change from baseline values.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Treatment
Number analyzed (Participants) | 15
fold change
  Day 7 | 18.60 (13.37)
  Month 3 | 4.04 (4.78)
Statistical Analysis 1: Comparison: Treatment; Test type: Other; A paired t-test was performed for skin lab measurement and biopsies

ADVERSE EVENTS:
Time Frame: 6 Months
Groups:
- Treatment: All patients will undergo treatment with Profound system device (microneedles and thermal heat to stimulate neocollagenesis). Using the radiofrequency and temperature setting within the FDA approved limits (460 +/- 5kHz and 65-75°C +/- 1°C), patients will be treated one time over the entire suprapatellar region bilaterally and followed for a 6 month period. The acute effect of the radiofrequency application will be determined by subjective and objective analysis using standard, close-up, 3D, cross-polarized, high resolution ultrasound, optical coherence tomography, transepidermal water loss measurements, and/or BTC 2000 measurements.
  Biopsies will be taken using 0.33mm WellTech Rapid Core 0.33mm Biopsy Punch. Biopsies will allow investigators to correlate changes seen in skin measurements with histology and gene expression.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=15)
Tenderness (Skin and subcutaneous tissue disorders) | 1 (1) — Event reported at Day 7
Tingling Sensation (Skin and subcutaneous tissue disorders) | 1 — Event reported on Day 7
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Event reported on Day 7
Swelling on the knee (Skin and subcutaneous tissue disorders) | 2 (2) — Event reported on Day 7
Blistering (Skin and subcutaneous tissue disorders) | 1 (1) — Event reported at Day 7
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT03507036/Prot_004.pdf
  • Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT03507036/SAP_005.pdf